CLINICAL TRIAL: NCT02353611
Title: Safety and Efficacy of a Light-activated 6% Hydrogen Peroxide With Nitrogen-doped Titanium Dioxide Tooth Bleaching Agent
Brief Title: Safety and Efficacy of a 6% Hydrogen Peroxide Tooth Bleaching Agent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Javier Martín, Prof.Javier Martín, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRI-ODO 15/001
Record Dates: First submitted 2015-01-22; First posted 2015-02-03 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Tooth Bleaching
Keywords: tooth; bleaching
MeSH Terms: interventions — Hydrogen Peroxide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 6% bleaching agent (Experimental): One upper hemiarch will be bleached with 6% hydrogen peroxide with titanium oxide nanoparticles, activated by a led/laser hybrid light. Whitening compound will be mixed according to manufacturer's instructions and distributed uniformly over the buccal surface of the teeth of one upper hemiarch. In each bleaching session the gel will be applied twice for 12 minutes each and activated with continuous irradiance using the LED/laser light (Whitening Lase Plus-DMC Equipamentos, São Carlos, SP, Brazil). Three bleaching sessions will be completed with an interval of 7 days between them.
  Interventions: Other: 6% hydrogen peroxide
- 35% bleaching agent (Active Comparator): Together with the experimental agent application, the other upper hemiarch will be bleached with 35% hydrogen peroxide whitening compound. The compound will be mixed according to manufacturer's instructions and distributed uniformly over the buccal surface of the teeth of the corresponding hemiarch. The gel will be applied twice for 12 minutes each and irradiated using the LED/laser light (Whitening Lase Plus-DMC Equipamentos, São Carlos, SP, Brazil). Three bleaching sessions will be completed with an interval of 7 days between them.
  Interventions: Other: 35% hydrogen peroxide

INTERVENTIONS:
Other: 6% hydrogen peroxide
  Other Names: 6% bleaching gel
  Arms: 6% bleaching agent
Other: 35% hydrogen peroxide — conventional peroxide whitening compound acted like control
  Other Names: 35%
  Arms: 35% bleaching agent

SUMMARY:
Bleaching protocol In each session, volunteers received prophylaxis with pumice powder and water. Then, gingival tissue was protected using a light-cured resin gum barrier applied according to the manufacturer's instructions (Lase Protect - DMC, São Carlos, SP, Brazil). Both bleaching agents were prepared by mixing hydrogen peroxide and thickening compounds according to the manufacturer's instructions (with 3 peroxide drops for 1 drop of thickener). The resultant gels were distributed uniformly on the upper hemiarcade surfaces of the teeth. A total of 8 teeth between the first premolars were bleached for each patient. In each bleaching session, the bleaching gels were applied twice for 12 minutes each. In each application, the surface of the gel was light activated with continuous irradiance for 12 minutes using LED/laser light with a total power of 1800 mW (Whitening Lase Plus - DMC Equipamentos, São Carlos, SP, Brazil). Three bleaching sessions were completed for the patients, and the interval between sessions was 7 days

DETAILED DESCRIPTION:
This was a randomized, triple-blinded (patients, evaluator, and statistician), and split-mouth design (one hemiarcade was treated by 1 compound) following nonprobability sampling. The patients were invited to participate in the study through posters posted around the city or recruited from participants in other studies in the same department, who were contacted by email or phone.

A total of 131 patients were examined in a dental chair to check if they met the inclusion and exclusion criteria. The patients included in this study were over 18 years old and selected with the following inclusion criteria: anterior teeth without restorations, previous bleaching procedures, cervical lesions, or dental pain. Patients who were pregnant or lactating, had moderate or severe fluorosis, tetracycline stains, orthodontic treatment, periodontal disease, orofacial tumors, trauma, or tooth malformation, or were taking analgesic, anti-inflammatory, or antibiotic drugs were excluded.

Two trained operators (restorative dentistry professors) performed the bleaching treatments. A third participant that did not have contact with the patients was responsible for conducting the randomization. The allocation of the hemiarcade in the groups was performed by random drawing using Microsoft Excel 2010 (Microsoft, Redmond, Washington, USA) from coding assigned to each participant. There were two experimental groups: Group A acted as a control, and hydrogen peroxide whitening compound was applied at a concentration of 35% to the upper hemiarcade. Group B was the experimental group, in which the other upper hemiarcade was treated with 6% compound catalyzed by titanium oxide nanoparticles and activated by blue hybrid light and an infrared laser.

The distribution of the operators was made by block randomization. To ensure triple blinding, the following procedures were adopted: 1) labels, logos, packaging, and any other aspect that could identify the products were removed, and procedures and instruments were standardized; 2) the bleaching protocol was performed in a different room from where the evaluator examined the patients; 3) the randomization was alpha-numerically coded to ensure blinding of the research team; and 5) a statistician received data tabulated in code that did not allow for identification of the treatment applied to each group.

Sample size calculation The primary outcome of this study was the efficacy determined by color alteration (ΔE). Previous studies showed that the use of in-office bleaching agent containing 35% hydrogen peroxide (HP35) with or without LED/Laser light leads to a ΔE value of 7.0-2.0 after two bleaching sessions. In order to have an 80% chance of detecting significance at the level of 5%, and considering an increase in the primary outcome measure from 7 in the control group to 5 in the experimental group, a minimum of 16 participants would be required in each group. Due to a higher dropout rate in the last two clinical studies of our research group, we decided to add 80% more patients, which led to 30 patients in each group.

Bleaching protocol In each session, volunteers received prophylaxis with pumice powder and water. Then, gingival tissue was protected using a light-cured resin gum barrier applied according to the manufacturer's instructions (Lase Protect - DMC, São Carlos, SP, Brazil). Both bleaching agents were prepared by mixing hydrogen peroxide and thickening compounds according to the manufacturer's instructions (with 3 peroxide drops for 1 drop of thickener). The resultant gels were distributed uniformly on the upper hemiarcade surfaces of the teeth. A total of 8 teeth between the first premolars were bleached for each patient. In each bleaching session, the bleaching gels were applied twice for 12 minutes each. In each application, the surface of the gel was light activated with continuous irradiance for 12 minutes using LED/laser light with a total power of 1800 mW (Whitening Lase Plus - DMC Equipamentos, São Carlos, SP, Brazil). Three bleaching sessions were completed for the patients, and the interval between sessions was 7 days.

Efficacy evaluation (E) Objective evaluation Two calibrated evaluators (Kappa=0.85) were used to measure the tooth color for the baseline (T0), immediately after the first (T1), second (T2), and third sessions (T3), and one week (T4) and one month after the third session (T5). The color evaluation was obtained from an area of 6 mm located in the middle third of the labial surface of the left and right central incisors. To standardize this evaluation, an impression of the maxillary arch was taken to make a guide using high-putty silicone (Zetaplus, Zhermack, Badia Polesine, Rovigo, Italy). A window was created on the labial surface in the middle third of the central incisor using a device with well-formed borders and a 3-mm radius corresponding to the reflectance of the spectrophotometer (Vita EasyShade Compact, VITA Zahnfabrik, Bad Säckingen, Germany). The shade was determined using the obtained parameters L*, a*, and b*. The color alteration after each session was given by the differences between the values obtained at the session and the baseline (∆E). ∆E was calculated using the following formula: ΔE = [(ΔL*)2 + (Δa*)2 + (Δb*)2]1/2 .

Subjective evaluation For the subjective evaluation, the 16 tabs of the shade guide (Vita Classic, Vita Zahnfabrik) were arranged from the highest (B1) to the lowest (C4) value. Although this scale is not linear in the truest sense, we treated the changes as continuous with a linear ranking, as was done in several clinical trials of dental bleaching. Two calibrated evaluators (Kappa=0.85) recorded the shade of the upper central left and right incisors at baseline with the same periods as the objective evaluation.

We checked the color in the middle third area of the labial surface of the anterior central incisor according to the American Dental Association guidelines. We calculated the color changes from the beginning of the active phase through the individual recall times by the change in the number of shade guide units (ΔSGU), which occurred toward the lighter end of the value-oriented list of shade tabs. In the event that the operators disagreed on color matching, a consensus was reached prior to dismissing the patient.

Tooth sensitivity evaluation (S) Tooth sensitivity was characterized by the variables occurrence, intensity, and type. These data were obtained by self-completed form and clinical evaluation during the session and immediately by VAS (Visual Analogue Scale). For the VAS, we instructed the participants to place a line perpendicular to a 10-mm-long line with zero at one end indicating ''no TS'' and the other end indicating ''unbearable TS.'' The occurrence was analyzed according to whether sensitivity was reported. The intensity was measured at four levels according to a verbal scale: 1=none, 2=mild, 3=moderate, 4=considerable, and 5=severe. The volunteers were instructed to fill out a form for each bleaching session and for the following days between sessions in case of sensitivity in any of the bleached teeth at any time.

ELIGIBILITY:
Inclusion Criteria:

* Anterior teeth without restorations, previous bleaching procedures, cervical lesions, or dental pain

Exclusion Criteria:

* Pregnant or lactating,
* had moderate or severe fluorosis, tetracycline stains, orthodontic treatment, periodontal disease, orofacial tumors, trauma, or tooth malformation, or
* were taking analgesic, anti-inflammatory, or antibiotic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Efectiveness by color difference (using the spectrophotometer Vita Easy Shade) | 1 month and 9 month
  Shade will be determined using L*, a*, and b* parameters measured by Spectrophotometer at 1 and 9 month after bleaching. The color change (ΔE) will be determined by the differences between the values obtained at each checkpoint and the baseline measures using the formula: ΔE = [(ΔL*)2 + (Δa*)2 + (Δb*)2]1/2

CONTACTS AND LOCATIONS:
Overall Officials: Javier Martín, Principal Investigator — University of Chile; Eduardo Fernandez, Study Director — University of Chile

REFERENCES:
- [Background] Bortolatto JF, Pretel H, Floros MC, Luizzi AC, Dantas AA, Fernandez E, Moncada G, de Oliveira OB Jr. Low Concentration H(2)O(2)/TiO_N in Office Bleaching: A Randomized Clinical Trial. J Dent Res. 2014 Jul;93(7 Suppl):66S-71S. doi: 10.1177/0022034514537466. Epub 2014 May 27. PMID 24868014
- [Background] Martin J, Fernandez E, Bahamondes V, Werner A, Elphick K, Oliveira OB Jr, Moncada G. Dentin hypersensitivity after teeth bleaching with in-office systems. Randomized clinical trial. Am J Dent. 2013 Feb;26(1):10-4. PMID 23724543
- [Background] Moncada G, Sepulveda D, Elphick K, Contente M, Estay J, Bahamondes V, Fernandez E, Oliveira OB, Martin J. Effects of light activation, agent concentration, and tooth thickness on dental sensitivity after bleaching. Oper Dent. 2013 Sep-Oct;38(5):467-76. doi: 10.2341/12-335-C. Epub 2013 Feb 7. PMID 23391030
- [Derived] Bersezio C, Martin J, Angel P, Bottner J, Godoy I, Avalos F, Fernandez E. Teeth whitening with 6% hydrogen peroxide and its impact on quality of life: 2 years of follow-up. Odontology. 2019 Jan;107(1):118-125. doi: 10.1007/s10266-018-0372-3. Epub 2018 Jun 30. PMID 29961213